CLINICAL TRIAL: NCT05769361
Title: Effect of a 12-week Training Program With Unstable Devices on Strength and Dynamic Balance in Older Adults
Brief Title: Training Programs Effects on Strength and Balance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UNST2223
Record Dates: First submitted 2022-10-11; First posted 2023-03-15 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Fall

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind study: only the researchers doing the study know which treatment or intervention the participant is receiving until the study is over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unstable (UNST) (Experimental): 12-week training protocol with unstable devices, twice a week.
  Interventions: Behavioral: UNST
- Stable (ST) (Experimental): 12-week training protocol with stable devices, twice a week
  Interventions: Behavioral: ST
- Control (CTRL) (No Intervention): No administration of training protocols.

INTERVENTIONS:
Behavioral: UNST — Strength and balance training using different destabilizing devices
  Arms: Unstable (UNST)
Behavioral: ST — Strength and balance training over firm surfaces
  Arms: Stable (ST)

SUMMARY:
Ageing involves several physiological changes such as loss of muscle mass, muscle strength, and alteration of balance control mechanisms. Consequently, there is an increased fall risk that can lead the older adult to a reduced self-sufficiency in daily living activities. Investigating the role of different physical activities to counteract the age-related declines deserves attention. The present study aimed to evaluate the effects of two trainings performed with and without unstable devices, on dynamic balance control and lower limb strength compared to a control group that received no intervention.

DETAILED DESCRIPTION:
The a-priori power analysis calculation reported a total sample size of 51 participants. We decided to increase the sample size of approximatively 20% hypothesizing an increment of drop-outs due to the not completely solved COVID-19 pandemic at the time of the study.

In this single-blinded randomized controlled study, both intervention groups received 24 training sessions of 45 minutes each, twice a week for 12 weeks.The two intervention groups and the control group were tested at the baseline (T0), after six weeks (T1), and after twelve weeks (T2).

Subjects of the intervention groups had to complete at least 21 out of 24 training sessions. Moreover, all subjects had to complete all the assessments. Otherwise, they were completely excluded from the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* self-sufficiency in daily living activities;
* aged between 65 and 85 years.

Exclusion Criteria:

* non-corrected sight disorders
* neurological disorders
* regular assumption of drugs that can interfere with normal cognitive functioning
* pathologies that contraindicate physical activity practice

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Center of Pressure (CoP) Unit Path | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  From the center of pressure (CoP) trajectory the following parameter is calculated in the dynamic test:
  - The mean velocity of the CoP measured in cm∙s-1 (Unit Path) over a 2.5-second time window from the beginning of the perturbation;
Center of Pressure (CoP) Area95 | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  From the center of pressure (CoP) trajectory the following parameter is calculated in the dynamic test:
  - The area of the 95th percentile confidence ellipse of the CoP measured in cm2 (Area95) over a 2.5-second time window from the beginning of the perturbation.
Center of Pressure (CoP) First Peak | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  From the center of pressure (CoP) trajectory the following parameter is calculated in the dynamic test:
  - First peak (FP) as the difference in centimeters between the peak reached by the CoP displacement after the external perturbation and the mean value of the anterior-posterior CoP displacement before the perturbation.
Center of Pressure (CoP) Maximal Oscillation | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  From the center of pressure (CoP) trajectory the following parameter is calculated in the dynamic test:
  - Maximal oscillation of the CoP anterior-posterior displacement as the sum in centimeters of the absolute values of FP and the subsequent peak.
Center of Pressure (CoP) Post Perturbation Variability | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  From the center of pressure (CoP) trajectory the following parameter is calculated in the dynamic test:
  - The standard deviation (SD) of the CoP anterior-posterior displacement over a 2.5-second time window from the beginning of the perturbation as the post perturbation variability (PPV), measured in centimeters.
Lower limb isometric strength | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  Isometric quadriceps maximal strength (Newton) measured with an instrumented chair. Specifically, a load cell is placed perpendicular to the subject's shank and collects the force in Newton expressed by the subject while sitting on the chair. The knee angle during the maximal effort is fixed at 90 degrees.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) test | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  Stand up from a chair, walk at the preferred pace to a cone at 3 meters, turn around, and walk back to the chair to sit down. The outcome is the time measured in seconds to complete the test.
10-meter walking test | At baseline (t0), after six weeks (t1) and after 12 weeks (t2)
  Walking 20 meters in a straight line at the preferred speed. The outcome is the time measured in seconds to complete the distance from the 5th to the 15th meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizzato A, Bozzato M, Rotundo L, Zullo G, De Vito G, Paoli A, Marcolin G. Multimodal training protocols on unstable rather than stable surfaces better improve dynamic balance ability in older adults. Eur Rev Aging Phys Act. 2024 Jul 12;21(1):19. doi: 10.1186/s11556-024-00353-8. PMID 38997647